CLINICAL TRIAL: NCT04275817
Title: Cognitive Prefrail and Frailty, and Motoric Cognitive Risk Syndrome: Prevalence and Association With Incident Adverse Health Events in the Canadian Longitudinal Study on Aging
Brief Title: Cognitive Prefrail and Frailty, and Motoric Cognitive Risk Syndrome: Prevalence and Association With Incident Adverse Health Events
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-2183
Record Dates: First submitted 2020-01-20; First posted 2020-02-19 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Frailty; Motoric Cognitive Risk Syndrome; Cognitive-prefrailty
MeSH Terms: conditions — Frailty | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with prefrailty: This is defined as a co-existing prefrailty using the Fried criteria. Frailty defined by the CHS index as proposed by Fried et al. will be identified by the presence of ≥ 3 of the following 5 components: 1) Shrinking: unintentional weight loss of ≥ 5% between two assessments, 2) Weakness: a maximal grip strength in the lowest quintile stratified by body mass index quartile; 3) Poor energy: answer of "no" to the question "Do you feel full of energy?" from the 15-item Geriatric Depression Scale; 4) Slowness: average walk speed in the lowest quintile stratified by median standing height, and 5) Low physical activity level: PASE score in the lowest quintile. Participants with none of the above components will be considered to be vigorous and those with 1 or 2 components will be considered to be in a prefrail stage.
  Interventions: Other: Data collection
- Individuals with cognitive-prefrailty: A combination of prefrailty stage using Fried criteria and subjective cognitive impairment (SCI).
  The IANA/IAGG consensus defines cognitive frailty as CDR = 0.5 and frailty by the Fried criteria.
  In this study, an individual will be considered a CHI if they meet the following criteria: no history of dementia, no use of anti-dementia drugs, normal cognitive performance on cognitive tests and normal scores of ADL and IADL scales. Different participant subgroups will be identified: 1) Individuals will be classified as MCI if they meet the following criteria: Objective cognitive impairment (i.e., performance between 1.5 and 1.9 SDs below the age-appropriate mean) in one or two cognitive domains (i.e., episodic memory and/or executive function) and normal scores of ADL and IADL scales; 2) Individuals will be considered older adults with mild-stage major neurocognitive disorders
  Interventions: Other: Data collection
- Individuals with MCR: The diagnosis of MCR syndrome will be made following the criteria of Verghese et al. 5: a combination of subjective cognitive complaint, in particular of memory complaint, with the presence of an objective slow gait and the absence of dementia or mobility disability. MCR syndrome will be defined at baseline assessment and each year of follow-up period. Slow gait speed will be defined as gait speed that is one standard deviation (SD) or more below age-and sex-appropriate mean values established in the present cohort like in previous studies. The mean value and SD of female and male will be determined separately. Gait speed was determined from the 3-meter walking test using the best time of the two trials recorded and expressed as meters per second.
  Memory complaint used to define MCR syndrome was based on standardized memory loss question on the 15-item Geriatric Depression Scale (GDS; "Do you feel you have more problems with memory than most?").
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Telephone interview questionnaire, in-home face-to-face interview, and data from the Collection Site

SUMMARY:
We defined a new and early condition in the spectrum of cognitive frailty: the "cognitive-prefrailty" which is a combination of prefrailty stage and subjective cognitive impairment (SCI). This study aims to: (1) examine and compare the prevalence of cognitive-prefrailty, cognitive frailty and motoric cognitive risk syndrome (MCR) syndromes in participants of the Canadian Longitudinal Study of Aging (CLSA) using the (tracking and comprehensive) baseline assessment, (2) examine the association of cognitive-prefrailty, cognitive frailty and MCR syndromes with incident adverse health events using the information collected during the first CLSA 18-month follow-up, and (3) compare the criteria performances (i.e., sensitivity, specificity, positive predictive value, negative predictive value, area under receiver operating characteristic curve, positive and negative likelihood ratio) for incident adverse health events of the cognitive-prefrailty, cognitive frailty and MCR syndromes.

DETAILED DESCRIPTION:
Background Cognitive frailty is the simultaneous presence of both physical frailty and cognitive impairment, excluding concurrent dementia. This condition confers a greater risk of incident cognitive impairment and decline, dementia, falls and disabilities compared to either condition alone. Current definitions of co-existent frailty and cognitive impairment exist, including the International Academy on Nutrition and Aging (IANA) and the International Association of Gerontology and Geriatrics (IAGG) consensus for cognitive frailty. There is also an analogous construct known as the motoric cognitive risk syndrome (MCR) associating slow gait speed and subjective cognitive impairment (SCI). Current operational criteria identify individuals later in the trajectory of frailty and cognitive decline, which may be too late for effective interventions. We propose to define a new and early condition in the spectrum of Cognitive frailty known as "cognitive-prefrailty", which is a combination of prefrailty stage and SCI.

Overall objective This study aims to: 1) Examine and compare the prevalence of cognitive-prefrailty, cognitive frailty and motoric cognitive risk syndrome (MCR) syndromes in participants of the Canadian Longitudinal Study of Aging (CLSA) using the (tracking and comprehensive) baseline assessment, 2) Examine the association of cognitive-prefrailty, cognitive frailty and MCR syndromes with incident adverse health events using the information collected during the first CLSA 18-month follow-up, 3) Compare the criteria performances (i.e., sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), area under receiver operating characteristic curve, positive and negative likelihood ratio (LR)) for incident adverse health events of the cognitive-prefrailty, cognitive frailty and MCR syndromes.

Methods This study will use the database of the CLSA, which is population-based observational and prospective cohort study that assesses and follows the health condition of the Canadian population. All items of cognitive-prefrailty, cognitive frailty and MCR syndromes have been collected during the baseline assessment in the tracking and the comprehensive assessments. In addition, all information needed to determine incident adverse health events including falls and related injuries, depression, functional decline, motoric cognitive risk syndrome, cognitive decline and dementia has been also collected during the first 18-month follow-up period.

Anticipated results Prefrailty is an intermediate and potentially reversible stage between robust and frailty that occur upstream in the continuum of frailty and hence constitute more suitable targets for screening and early intervention in older adults.

ELIGIBILITY:
Inclusion Criteria:

1. participants of the CLSA with baseline assessment (tracking and comprehensive assessment) and first 18-month follow-up assessment
2. age > 50

Exclusion Criteria:

1. no information which may directly or indirectly determine the occurrence of incident adverse health events (falls and related injuries, depression, functional decline, motoric cognitive risk syndrome, cognitive decline and dementia)
2. age < 50 and demented LCSA participants if they meet the following criteria:

   1. History of dementia or Alzheimer's disease and/or use of anti-dementia drugs (i.e., Donepezil, Rivastigmine, Galentamine, regardless the dose taken)
   2. Objective cognitive impairment (i.e., performance ≥2 SDs below the age-appropriate mean) in two cognitive domains (i.e., episodic memory and executive function) and abnormal scores on the ADL and IADL scales

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals eligible for this study will be the participants of the CLSA
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive-prefrailty | 1 day
  Defined as frailty and subjective cognitive impairment combined. Frailty (as proposed by Fried et al.) will be identified by the presence of ≥ 3 of the 5 components: 1) unintentional weight loss, 2) Weakness (maximal grip strength); 3) Poor energy (answer of "no" to the question "Do you feel full of energy?" from the 15-item Geriatric Depression Scale); 4) Slowness as identified by an average walk speed, and 5) Low physical activity level. Participants with none of the above components will be considered to be vigorous and those with 1 or 2 components will be considered to be in a prefrail stage.
  SCI will be defined using a proxy for subjective cognitive complaint (i.e. memory complaint) based on standardized memory loss question on the 15-item Geriatric Depression Scale (GDS; "Do you feel you have more problems with memory than most?").

SECONDARY OUTCOMES:
Falls | 12 months
  Number of falls
Depression | 1 day
  10 items from the Center for Epidemiological Studies' Short Depression Scale (CES-D) score ≥10
Activities daily living (ADL) | 1 day
  ADL score out of 6. Where a score of 3-5 is indicative of mild stages of neurocognitive disorders.
Motoric Cognitive Risk | 1 day
  Defined as having subjective cognitive complaint and slow walking speed (subjective cognitive complaint will be defined using the variable trouble concentrating or the self-reported memory problem, and slow walking speed will be defined as walking speed one standard deviation (SD) below the average of the cohort using the information of modules psychological health and physical health)

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada